CLINICAL TRIAL: NCT03223883
Title: Curcumin Supplementation for Improving Vascular and Cognitive Function in Chronic Kidney Disease
Brief Title: Curcumin and Vascular and Cognitive Function in Patients With Chronic Kidney Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Diana Jalal (Other)
Collaborators: University of Colorado, Boulder (Other); Stanford University (Other); University of Colorado, Denver (Other)
Responsible Party: Sponsor-Investigator, Diana Jalal, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201710769
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Chronic Kidney Diseases; Cognitive Decline
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cognitive Dysfunction | interventions — Curcumin

STUDY DESIGN:
Intervention Model Description: Randomized Double-Blind Placebo-Controlled Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patient, providers, and the investigative team will all be blinded to the randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Curcumin (Experimental): Patients will receive curcumin (Lonvida) 2000 mg PO once a day
  Interventions: Drug: Curcumin
- Placebo (Placebo Comparator): Patients will receive placebo pill identical in appearance and taste to the supplement
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Curcumin — Oral supplement for 12 months
  Other Names: Longvida
  Arms: Curcumin
Other: Placebo — Oral placebo for 12 months
  Arms: Placebo

SUMMARY:
The proposed research is clinical study evaluating the therapeutic benefits of curcumin on vascular function in patients with chronic kidney disease (CKD). The study aims to establish that curcumin will improve endothelial function and reduce large artery stiffness by reducing oxidative stress and in conjunction with lowering markers of inflammation and oxidative stress. In addition, the study will evaluate the potential benefit of curcumin on cognitive function in patients with CKD.

DETAILED DESCRIPTION:
Patients with chronic kidney disease (CKD) are at increased risk of death from cardiovascular disease (CVD). Inflammation, oxidative stress and vascular dysfunction (impaired endothelial function and increased large elastic artery stiffness), are highly prevalent in CKD and contribute to the high incidence of CVD in this patient population. In addition, patients with CKD suffer from high rates of cognitive decline for which we lack effective therapies. Thus, therapeutic interventions targeting inflammation, oxidative stress, vascular dysfunction, and cognitive impairment in CKD are a biomedical priority.

Curcumin is a natural polyphenol with anti-inflammatory and antioxidant characteristics. It is safe and widely-available. Preliminary data in old mice and healthy middle-aged (MA)/older adult humans indicate that curcumin administration improves endothelial dysfunction and large artery stiffness by reducing oxidative stress and inflammation. Additionally, 12 weeks of curcumin supplementation improves episodic memory in MA/older adults.

The primary goal of this R01 application is to extend previous findings in healthy MA/older adults to patients with CKD, a growing clinical population with extensive baseline vascular dysfunction and cognitive impairment who presently have few treatment options. The hypothesis is that curcumin improves vascular endothelial function and large elastic artery stiffness in MA/older adults with stage IIIb and IV CKD (estimated GFR 15-45 mL/min/1.73m2). The possible mechanisms by which curcumin improves vascular function will be evaluated as well as whether curcumin improves cognitive function in these patients.

Specific aim 1a will determine if 12 months of curcumin supplementation will improve brachial artery-flow mediated dilation (BA-FMD) (endothelial function) and aortic pulse wave velocity (aPWV) (arterial stiffness) compared to placebo (randomized placebo-controlled double-blind study). Specific aim 1b will evaluate whether the curcumin-induced improvements in BA-FMD and aPWV are mediated by reduced oxidative stress, and will evaluate the effects of curcumin on systemic and endothelial cell markers of inflammation and oxidative stress. Importantly, specific aim 2 will evaluate the effects of curcumin supplementation on cognitive function, an important complication of CKD, using the NIH Cognitive Toolbox Battery.

ELIGIBILITY:
Inclusion Criteria:

* CKD stage IIIB and IV
* BMI<35 kg/m2
* Able to give informed consent

Exclusion Criteria:

* Consuming a diet rich in curcumin or taking curcumin supplements in the past 12 months
* Life expectancy <1 year
* Pregnant, breastfeeding, or unwilling to use adequate birth control
* Uncontrolled hypertension
* Severe liver disease
* Severe congestive heart failure
* Hospitalization within the last 3 months
* Active infection or antibiotic therapy
* Immunosuppressive therapy within the last year

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Jalal, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited between June 2018 and February 2022 from the Renal Clinics at the University of Iowa Hospital and Clinics (UIHC) and the Iowa City Veterans Affairs Health Care System (VA HCS). All procedures were approved by the University of Iowa and the Iowa City VA HCS Institutional Review Boards and conducted in accordance with the Declaration of Helsinki. All participants provided written documentation of the informed consent process before study participation.
Period: Overall Study
Arm/Group | Curcumin | Placebo
Started | 45 | 43
Completed | 37 | 38
Not Completed | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Curcumin | Placebo | Total
Number analyzed (Participants) | 45 | 43 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (8) | 65 (8) | 66 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 35 | 31 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 45 | 42 | 87
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 41 | 40 | 81
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 45 | 43 | 88
Brachial artery flow-mediated dilation [Median (Inter-Quartile Range); unit: % change] | 2.8 [1.7 to 4.2] | 2.6 [1.5 to 3.3] | 2.7 [1.6 to 3.7]

OUTCOME MEASURES:

1. Primary Outcome: Change in Vascular Endothelial Function at 12 Months
Description: Brachial artery flow-mediated dilation, changed in diameter in brachial artery in response to shear stress
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: %change
Arm/Group | Curcumin | Placebo
Number analyzed (Participants) | 37 | 38
%change | -0.1 [-1.5 to 1.5] | -0.7 [-2.1 to 1.1]

2. Secondary Outcome: Large Artery Stiffness
Description: Aortic pulse wave velocity
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Curcumin | Placebo
Number analyzed (Participants) | 37 | 38
m/s | 0.28 (2.4) | 0.36 (4.2)

3. Secondary Outcome: Cognitive Function
Description: NIH toolbox battery- Executive Function Age-Corrected Standard Score is reported (T-score): This score compares the score of the test-taker to those in the NIH Toolbox nationally representative normative sample at the same age, where a score of 100 indicates performance that was at the national average for the test-taking participant's age. Age-corrected standard scores were derived separately for children (ages 3-17) and adults (ages 18-85). A score of 115 or 85, for example, would indicate that the participant's performance is 1 SD above or below the national average, respectively, when compared with like-aged participants. Higher scores indicate better performance.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: age-adjusted T-score
Arm/Group | Curcumin | Placebo
Number analyzed (Participants) | 37 | 38
age-adjusted T-score | 2.62 (9) | 2.25 (9.5)

ADVERSE EVENTS:
Time Frame: 12 MONTHS
Arm/Group | Curcumin | Placebo
All-Cause Mortality (participants affected / at risk) | 1/45 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/43
Other Adverse Events (participants affected / at risk) | 27/45 | 21/43
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Curcumin (N=45) | Placebo (N=43)
Nausea (Gastrointestinal disorders) | 7 | 6
Vomiting (Gastrointestinal disorders) | 4 | 6
Abdominal PAIN (Gastrointestinal disorders) | 6 | 2
Dizziness (General disorders) | 10 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-08-19): https://cdn.clinicaltrials.gov/large-docs/83/NCT03223883/Prot_003.pdf
  • Statistical Analysis Plan (2024-08-19): https://cdn.clinicaltrials.gov/large-docs/83/NCT03223883/SAP_004.pdf
  • Informed Consent Form (2022-08-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT03223883/ICF_002.pdf